CLINICAL TRIAL: NCT05852236
Title: The Effect of Pressure Wound Care Package on O.R. Pressure Wound Development
Brief Title: The Effect of Pressure Wound Care Package on the Development of Operating Room Pressure Wound in Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehitkamil Devlet Hastanesi (Other)
Responsible Party: Principal Investigator, Hatice Eğilmez, Nurse, RN, Sehitkamil Devlet Hastanesi
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: ŞehitkamilDH275002727
Record Dates: First submitted 2023-04-04; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pressure Injury; Orthopedic Surgery
Keywords: orthopedic surgery; pressure injury; care bundle; pain; fear of falling; comfort
MeSH Terms: conditions — Pressure Ulcer; Pain

STUDY DESIGN:
Masking Description: Non-Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): The standard care of the clinic was applied to the control group.
  Interventions: Other: Assigned Interventions
- Study Group (Experimental): The pressure ulcer care package developed for this study was applied to the study group.
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Pressure ulcer care package application.

SUMMARY:
SUMMARY In a non-randomised (quasi-experimental) clinical study, it was aimed to determine the effect of the care package applied in the early postoperative period on operating theatre pressure sores, pain, fear of falling and comfort in patients undergoing orthopaedic surgery. In the study, the care bundle for pressure injuries was prepared in accordance with the clinical guidelines and was applied to the patients in the study group. This study was conducted in the orthopaedics and traumatology clinic of a public hospital in the Southeastern Anatolia Region of Turkey.

DETAILED DESCRIPTION:
Medhod:Patients in the control group underwent routine practice of the clinic and this group was observed for 199 days. The care bundle for pressure injuries developed within the scope of the research was not applied. In the study group, in addition to routine clinical practice, the care bundle for pressure injuries developed for this study was applied for 105 days. Since the pressure ulcer originating from the operating room was seen until the 48th-72nd hour, the evaluations and interventions within the scope of the study were performed for three days, considering the operation day as the zeroth day for the control and study groups. A total of 190 patients, 122 in the control group and 68 in the study group, were included in the study.

The care bundle consisted of "skin care, positioning, early mobilization, nutrition, and fluid intake" interventions. In the study, first, the data of the control group and then the data of the study group were collected.

Data Collection Tools: The Patient Descriptive Information Form consists of sociodemographic data. The 3S OR Pressure Injury Risk Assessment Scale was used to identify patients at risk of developing OR pressure ulcers. Visual Analogue Scale was used to evaluate pain perception. The Visual Analog Scale was used to determine the fear of falling. General Comfort Questionnaire-Short Form was used to determine the comfort level. The National Pressure Ulcer Advisory Panel (NPUAP) 2016 Pressure Injury Staging System was used to assess and stage pressure ulcer development. Pressure Injury Areas and Stages Follow-up Registration Form; The form in which the pressure ulcer development status is recorded.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older

* Orthopaedics and traumatology department
* Those who have undergone general or spinal anaesthesia
* No history of surgery in the last month
* Without any communication problems
* 3S Patients with a score of 18 and above on the Operating Theatre Pressure Wound Risk Assessment Scale
* Patients admitted to the emergency clinic, whose trauma-related surgery is planned within 24 hours from the emergency clinic
* Admission to the orthopaedics and traumatology clinic within maximum 24 hours from the day of surgery planned as elective surgery
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* I'm the one whose surgery was cancelled
* Those who have undergone local or regional anaesthesia
* Patients referred to the intensive care unit after surgery
* Patients who wanted to leave the study after volunteering were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The effect of pressure ulcer care package on the incidence of pressure ulcers in patients | Implementation Time: 3.5 Month
  In this study, it was seen that the pressure ulcer care package applied to the study group contributed positively to the change in the incidence rate of pressure ulcers.
The effect of pressure ulcer care package on pain perception in patients | Implementation Time: 3.5 Month
  In this study, it was seen that the pressure ulcer care package applied to the study group made positive contributions to the change of pain level.
  Visual Analog Scale was used to evaluate the level of pain. The score obtained from the scale ranges from one to ten. The higher the score, the higher the level of pain.
The effect of pressure ulcer care package on fear of falling in patients | Implementation Time: 3.5 Month
  In this study, the pressure ulcer care package applied to the study group changed the fear of falling in patients.
  Visual Analogue Scale was used to obtain numerical data in the assessment of fear of falling. The score obtained from the scale ranges from one to ten. The higher the score, the greater the fear of falling.
The effect of pressure ulcer care package on comfort in patients | Implementation Time: 3.5 Month
  In this study, the pressure ulcer care package applied to the study group changed the comfort of the patients.
  The comfort level of the patients was determined by using the short form of the comfort scale. As the score obtained from the scale increases, the level of comfort increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla YAVA, PhD, Study Director — Prefessor
Locations (1):
- Şehitkamil Devlet Hastanesi, Gaziantep, Turkey (Türkiye)